CLINICAL TRIAL: NCT02977949
Title: The Effects of Seasonal Changes in Osteoporosis Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Toshihiko Kono (Other)
Responsible Party: Sponsor-Investigator, Toshihiko Kono, Head of Hospital, Tomidahama Hospital
Organization: Tomidahama Hospital (Other)
Other Study IDs: TH 05-2
Record Dates: First submitted 2016-11-23; First posted 2016-11-30 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Selective Estrogen Receptor Modulator (SERM)
Keywords: SERM; Season; Variation; Vitamin D
MeSH Terms: interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months

INTERVENTIONS:
Drug: Raloxifene

SUMMARY:
There are few reports concerning to the seasonal variation of osteoporosis treatment. In this study, we plan to compare clinical efficacy and safety by seasons.

DETAILED DESCRIPTION:
Vitamin D insufficiency is common in many countries. Vitamin D insufficiency is associated with osteoporosis and the responses to osteoporosis treatment. 25-hydroxyvitamin D (25OHD) is considered to be the best estimate of body stores of vitamin D and the seasonal variation of 25OHD is well known. But there are few reports concerning to the seasonal variation of osteoporosis treatment. In this study, we plan to compare clinical efficacy and safety by seasons in patients treated by raloxifene.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women

Exclusion Criteria:

* Patients who could not use SERM

Ages: 45 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Osteoporosis patients using raloxifene more for two years.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2012-01; Primary Completion 2018-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Effects of raloxifene on bone mineral density in postmenopausal osteoporosis. | Up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Rui Niimi, MD, Study Director — Tomidahama Hospital
Locations (1):
- Tomidahama Hospital, Yokkaichi, Mie-ken, Japan